CLINICAL TRIAL: NCT00393458
Title: A 52-week Treatment, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Indacaterol (300 and 600 µg Once Daily) in Patients With Chronic Obstructive Pulmonary Disease, Using Formoterol (12 µg Twice Daily) as an Active Control
Brief Title: Efficacy, Safety, and Tolerability of Once Daily Indacaterol in Chronic Obstructive Pulmonary Disease (COPD) Using Formoterol Twice Daily as Active Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2334
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol; long-acting β2 agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Indacaterol 300 μg plus placebo to formoterol (Experimental): Patients inhaled indacaterol 300 μg once daily via a single-dose dry-powder inhaler (SDDPI), placebo to indacaterol once daily via a SDDPI, and placebo to formoterol twice daily via the manufacturer's proprietary inhalation device (Aerolizer®). Indacaterol, placebo to indacaterol, and placebo to formoterol were taken in the morning between 8:00 and 10:00 AM; placebo to formoterol was taken again 12 hours later in the evening between 8:00 and 10:00 PM. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to formoterol
- Indacaterol 600 μg plus placebo to formoterol (Experimental): Patients inhaled indacaterol 600 μg (two 300 μg capsules) once daily via single-dose dry-powder inhalers (SDDPI) plus placebo to formoterol twice daily via the manufacturer's proprietary inhalation device (Aerolizer®). Indacaterol and placebo to formoterol were taken in the morning between 8:00 and 10:00 AM; placebo to formoterol was taken again 12 hours later in the evening between 8:00 and 10:00 PM. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to formoterol
- Formoterol 12 μg plus placebo to indacaterol (Active Comparator): Patients inhaled formoterol 12 μg twice daily via the manufacturer's proprietary inhalation device (Aerolizer®) plus placebo to indacaterol once daily via a single-dose dry-powder inhaler (SDDPI). Formoterol and placebo to indacaterol were taken in the morning between 8:00 and 10:00 AM; formoterol was taken again 12 hours later in the evening between 8:00 and 10:00 PM. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Formoterol; Drug: Placebo to indacaterol
- Placebo to indacaterol plus placebo to formoterol (Placebo Comparator): Patients inhaled placebo to indacaterol once daily via a single-dose dry-powder inhaler (SDDPI) plus placebo to formoterol twice daily via the manufacturer's proprietary inhalation device (Aerolizer®). Placebo to indacaterol and placebo to formoterol were taken in the morning between 8:00 and 10:00 AM; placebo to formoterol was taken again 12 hours later in the evening between 8:00 and 10:00 PM. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol; Drug: Placebo to formoterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol was supplied in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Indacaterol 300 μg plus placebo to formoterol; Indacaterol 600 μg plus placebo to formoterol
Drug: Formoterol — Formoterol was supplied in powder-filled capsules with the manufacturer's proprietary inhalation device (Aerolizer®).
  Arms: Formoterol 12 μg plus placebo to indacaterol
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder-filled capsules with a single-dose dry-powder inhaler (SDDPI).
  Arms: Formoterol 12 μg plus placebo to indacaterol; Placebo to indacaterol plus placebo to formoterol
Drug: Placebo to formoterol — Placebo to formoterol was supplied in powder-filled capsules with the manufacturer's proprietary inhalation device (Aerolizer®).
  Arms: Indacaterol 300 μg plus placebo to formoterol; Indacaterol 600 μg plus placebo to formoterol; Placebo to indacaterol plus placebo to formoterol

SUMMARY:
This study was designed to assess the efficacy and long-term safety of 300 and 600 µg doses of indacaterol when delivered via a single-dose dry-powder inhaler (SDDPI) in patients with chronic obstructive pulmonary disease (COPD). Patients were randomized to receive either indacaterol 300 µg once daily, indacaterol 600 µg once daily, formoterol 12 µg twice daily, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ≥ 40 years, with a diagnosis of chronic obstructive pulmonary disease (COPD) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines 2005 and:

  1. Smoking history of at least 20 pack years
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (forced volume capacity) < 70% (Post refers to within 30 minutes after inhalation of 400 μg of salbutamol)

     Exclusion Criteria:
* Patients who were hospitalized for a COPD exacerbation in the 6 weeks prior to screening.
* Patients who had a respiratory tract infection within 6 weeks prior to screening.
* Patients with concomitant pulmonary disease.
* Patients with a history of asthma.
* Patients with diabetes type I or uncontrolled diabetes type II.
* Any patient with lung cancer or a history of lung cancer.
* Patients with a history of certain cardiovascular co-morbid conditions.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1732 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Investigator Site, Principal Investigator — Novartis
Locations (183):
- Argentina (5):
  - Novartis Investigator Site, Buenos Aires
  - Novartis, Buenos Aires
  - Novartis Investigator Site, Mendoza
  - Novartis Investigator Site, San Miguel
  - Novartis Investigator Site, Santa Fe
- Chile (3):
  - Novartis Investigator Site, Rancagua
  - Novartis, Santiago
  - Novartis Investigator Site, Viña del Mar
- Colombia (3):
  - Novartis Investigator Site, Barranquilla
  - Novartis, Bogotá
  - Novartis Investigator Site, Medellín
- Czechia (7):
  - Novartis Investigator Site, Cvikov
  - Novartis Investigator Site, Kyjov
  - Novartis Investigator Site, Ostrava Poruba
  - Novartis Investigator Site, Pardubice
  - Novartis, Prague
  - Novartis Investigator Site, Tábor
  - Novartis Investigator Site, Žatec
- Denmark (6):
  - Novartis Investigator Site, Aarhus
  - Novartis, Copenhagen
  - Novartis Investigator Site, Hellerup
  - Novartis Investigator Site, Hvidovre
  - Novartis Investigator Site, Molleparkvej
  - Novartis Investigator Site, Odense
- Ecuador (3):
  - Novartis Investigator Site, Guayaquil
  - Novartis Investigator Site, Quito
  - Novartis, Quito
- Egypt (4):
  - Novartis Investigator Site, Alexandria
  - Novartis Investigator Site, Asyut
  - Novartis Investigator Site, Cairo
  - Novartis, Cairo
- Estonia (2):
  - Novartis Investigator Site, Tallinn
  - Novartis, Tartu
- France (12):
  - Novartis Investigator Site, Beuvry
  - Novartis Investigator Site, Chamalières
  - Novartis Investigator Site, Férolles-Attilly
  - Novartis Investigator Site, Grasse
  - Novartis Investigator Site, Marseille
  - Novartis Investigator Site, Montpellier
  - Novartis Investigator Site, Nice
  - Novartis Investigator Site, Nîmes
  - Novartis Investigator Site, Paris
  - Novartis Investigator Site, Perpignan
  - Novartis Investigator Site, Pessac
  - Novartis Investigator Site, Strasbourg
- Germany (38):
  - Novartis Investigator Site, Augsburg
  - Novartis Investigator Site, Bad Segeberg
  - Novartis Investigator Site, Bad Wörishofen
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bielefeld
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Borstel
  - Novartis Investigator Site, Darmstadt
  - Novartis Investigator Site, Dortmund
  - Novartis Investigator Site, Erfurt
  - Novartis Investigator Site, Forchheim
  - Novartis Investigator Site, Frankfurt
  - Novartis Investigator Site, Gauting
  - Novartis Investigator Site, Geesthacht
  - Novartis Investigator Site, Gelsenkirchen
  - Novartis Investigator Site, Großhansdorf
  - Novartis Investigator Site, Gummersbach
  - Novartis Investigator Site, Hagen
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Ilvesheim
  - Novartis Investigator Site, Kassel
  - Novartis Investigator Site, Kiel
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Lübeck
  - Novartis Investigator Site, Lüdenscheid
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Marburg
  - Novartis Investigator Site, München
  - Novartis Investigator Site, Neumünster
  - Novartis, Nuremberg
  - Novartis Investigator Site, Oschersleben
  - Novartis Investigator Site, Rüdersdorf
  - Novartis Investigator Site, Schönefeld
  - Novartis Investigator Site, Strausberg
  - Novartis Investigator Site, Witten
  - Novartis Investigator Site, Wuppertal
- Hungary (6):
  - Novartis Investigator Site, Budapest
  - Novartis, Budapest
  - Novartis Investigator Site, Deszk
  - Novartis Investigator Site, Mátraháza
  - Novartis Investigator Site, Mosdós
  - Novartis Investigator Site, Sopron
- Israel (4):
  - Novartis Investigator Site, Jerusalem
  - Novartis, Petah Tikva
  - Novartis Investigator Site, Rehovot
  - Novartis Investigator Site, Tel Litwinsky
- Italy (11):
  - Novartis Investigator Site, Ancona
  - Novartis Investigator Site, Catania
  - Novartis Investigator Site, Ferrara
  - Novartis Investigator Site, Florence
  - Novartis Investigator Site, Foggia
  - Novartis Investigator Site, Genova
  - Novartis Investigator Site, Milan
  - Novartis, Milan
  - Novartis Investigator Site, Pisa
  - Novartis Investigator Site, Roma
  - Novartis Investigator Site, Siena
- Latvia (4):
  - Novartis Investigator Site, Daugavpils
  - Novartis Investigator Site, Jēkabpils
  - Novartis Investigator Site, Riga
  - Novartis, Riga
- Lithuania (5):
  - Novartis Investigator Site, Alytus
  - Novartis Investigator Site, Kaunas
  - Novartis, Kaunas
  - Novartis Investigator Site, Klaipėda
  - Novartis Investigator Site, Vilnius
- Netherlands (15):
  - Novartis Investigator Site, Almelo
  - Novartis Investigator Site, Amersfoort
  - Novartis, Arnhem
  - Novartis Investigator Site, Breda
  - Novartis Investigator Site, Ede
  - Novartis Investigator Site, Eindhoven
  - Novartis Investigator Site, Harderwijk
  - Novartis Investigator Site, Helmond
  - Novartis Investigator Site, Hengelo
  - Novartis Investigator Site, Hoorn
  - Novartis Investigator Site, Leeuwarden
  - Novartis Investigator Site, Rotterdam
  - Novartis Investigator Site, Sneek
  - Novartis Investigator Site, Veldhoven
  - Novartis Investigator Site, Zutphen
- Peru (2):
  - Novartis Investigator Site, Lima
  - Novartis, Lima
- Romania (4):
  - Novartis, Bucharest
  - Novartis Investigator Site, Cluj-Napoca
  - Novartis Investigator Site, Iași
  - Novartis Investigator Site, Timișoara
- Russia (6):
  - Novartis Investigator Site, Kazan'
  - Novartis Investigator Site, Moscow
  - Novartis, Moscow
  - Novartis Investigator Site, Saint Petersburg
  - Novartis Investigator Site, Samara
  - Novartis Investigator Site, Yekaterinburg
- Slovakia (5):
  - Novartis Investigator Site, Banská Bystrica
  - Novartis Investigator Site, Bratislava
  - Novartis, Bratislava
  - Novartis Investigator Site, Košice
  - Novartis Investigator Site, Partizánske
- South Korea (5):
  - Novartis Investigator Site, Kyunggi
  - Novartis Investigator Site, Seoul
  - Novartis, Seoul
  - Novartis Investigator Site, Suwon
  - Novartis Investigator Site, Uijeongbu-si
- Spain (11):
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis, Barcelona
  - Novartis Investigator Site, Begonte
  - Novartis Investigator Site, Cáceres
  - Novartis Investigative Site, Madrid
  - Novartis Investigator Site, Mataró
  - Novartis Investigator Site, Petrel
  - Novartis Investigator Site, Ponferrada
  - Novartis Investigator Site, Terrassa
  - Novartis Investigator Site, Valencia
- Switzerland (5):
  - Novartis Investigator Site, Aarau
  - Novartis Investigator Site, Basel
  - Novartis Investigator Site, Locarno
  - Novartis Investigator Site, Münchenstein
  - Novartis Investigator Site, Zurich
- Turkey (Türkiye) (6):
  - Novartis Investigator Site, Ankara
  - Novartis Investigator Site, Bursa
  - Novartis, Istanbul
  - Novartis Investigator Site, Izmir
  - Novartis Investigator Site, Mersin
  - Novartis Investigator Site, Yenişehir
- United Kingdom (11):
  - Novartis Investigator Site, Belfast
  - Novartis Investigator Site, Bexhill-on-Sea
  - Novartis Investigator Site, Blackpool
  - Novartis Investigator Site, Chertsey
  - Novartis Investigator Site, Glasgow
  - Novartis Investigator Site, Leicester
  - Novartis Investigator Site, London
  - Novartis Investigator Site, Manchester
  - Novartis Investigator Site, Newcastle upon Tyne
  - Novartis Investigator Site, Slough
  - Novartis Investigator Site, Swansea

REFERENCES:
- [Derived] Jones PW, Donohue JF, Nedelman J, Pascoe S, Pinault G, Lassen C. Correlating changes in lung function with patient outcomes in chronic obstructive pulmonary disease: a pooled analysis. Respir Res. 2011 Dec 29;12(1):161. doi: 10.1186/1465-9921-12-161. PMID 22206353
- [Derived] Bleecker ER, Siler T, Owen R, Kramer B. Bronchodilator efficacy and safety of indacaterol 150 mug once daily in patients with COPD: an analysis of pooled data. Int J Chron Obstruct Pulmon Dis. 2011;6:431-8. doi: 10.2147/COPD.S21073. Epub 2011 Aug 18. PMID 22003288
- [Derived] Jones PW, Mahler DA, Gale R, Owen R, Kramer B. Profiling the effects of indacaterol on dyspnoea and health status in patients with COPD. Respir Med. 2011 Jun;105(6):892-9. doi: 10.1016/j.rmed.2011.02.013. Epub 2011 Mar 11. PMID 21397482
- [Derived] Worth H, Chung KF, Felser JM, Hu H, Rueegg P. Cardio- and cerebrovascular safety of indacaterol vs formoterol, salmeterol, tiotropium and placebo in COPD. Respir Med. 2011 Apr;105(4):571-9. doi: 10.1016/j.rmed.2010.11.027. Epub 2011 Jan 11. PMID 21227674
- [Derived] Dahl R, Chung KF, Buhl R, Magnussen H, Nonikov V, Jack D, Bleasdale P, Owen R, Higgins M, Kramer B; INVOLVE (INdacaterol: Value in COPD: Longer Term Validation of Efficacy and Safety) Study Investigators. Efficacy of a new once-daily long-acting inhaled beta2-agonist indacaterol versus twice-daily formoterol in COPD. Thorax. 2010 Jun;65(6):473-9. doi: 10.1136/thx.2009.125435. PMID 20522841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 300 μg Plus Placebo to Formoterol | Indacaterol 600 μg Plus Placebo to Formoterol | Formoterol 12 μg Plus Placebo to Indacaterol | Placebo to Indacaterol Plus Placebo to Formoterol
Started | 437 | 428 | 435 | 432
Exposed to Study Medication or Placebo | 437 | 425 | 434 | 432
Completed | 338 | 326 | 323 | 295
Not Completed | 99 | 102 | 112 | 137
Not completed — Adverse Event | 35 | 24 | 40 | 35
Not completed — Subject withdrew consent | 27 | 40 | 33 | 50
Not completed — Unsatisfactory therapeutic effect | 12 | 9 | 12 | 30
Not completed — Protocol deviation | 11 | 11 | 11 | 10
Not completed — Administrative problems | 7 | 8 | 5 | 2
Not completed — Lost to Follow-up | 5 | 6 | 5 | 3
Not completed — Abnormal laboratory value(s) | 1 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 5 | 5
Not completed — Abnormal test procedure result(s) | 0 | 1 | 1 | 2
Not completed — Subject no longer requires study drug | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 300 μg Plus Placebo to Formoterol | Indacaterol 600 μg Plus Placebo to Formoterol | Formoterol 12 μg Plus Placebo to Indacaterol | Placebo to Indacaterol Plus Placebo to Formoterol | Total
Number analyzed (Participants) | 437 | 425 | 434 | 432 | 1728
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are based on all subjects in the safety population, which includes all patients who received at least 1 dose of study drug. Three patients in the indacaterol 600 μg plus placebo to formoterol and one patient in the formoterol 12 μg plus placebo to indacaterol group were not exposed to any study treatment.
  years | 63.9 (8.57) | 62.9 (8.74) | 63.6 (8.49) | 63.2 (8.28) | 63.4 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 98 | 86 | 80 | 350
  Male | 351 | 327 | 348 | 352 | 1378

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12 + 1 Day, Day 85
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: Week 12 + 1 day, Day 85
Population: Modified intent-to-treat (ITT) population: All randomized patients who received at least 1 dose of study drug, excluding patients from a number of centers.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg Plus Placebo to Formoterol | Indacaterol 600 μg Plus Placebo to Formoterol | Formoterol 12 μg Plus Placebo to Indacaterol | Placebo to Indacaterol Plus Placebo to Formoterol
Number analyzed (Participants) | 389 | 374 | 379 | 371
Liters | 1.48 (0.012) | 1.48 (0.013) | 1.38 (0.013) | 1.31 (0.013)

2. Secondary Outcome: Percentage of Days of Poor Control During 52 Weeks of Treatment
Description: Percentage of days of poor control was defined as the number of days in the patient diary with a score ≥ 2 (scale of 0-3, a higher number means more severe symptoms) for at least 2 of 5 symptoms (cough, wheeze, production of sputum, color of sputum, breathlessness) over 52 weeks divided by the number of evaluable days (days with ≥ 2 symptoms with scores). The analysis included baseline percentage of days of poor control, FEV1 pre-dose and 30 minutes post-dose of salbutamol/albuterol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: Baseline to end of study (Week 52)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol 300 μg Plus Placebo to Formoterol | Indacaterol 600 μg Plus Placebo to Formoterol | Formoterol 12 μg Plus Placebo to Indacaterol | Placebo to Indacaterol Plus Placebo to Formoterol
Number analyzed (Participants) | 386 | 370 | 377 | 366
Percentage of days | 33.6 (1.43) | 30.0 (1.46) | 33.5 (1.45) | 38.3 (1.47)

ADVERSE EVENTS:
Time Frame: Safety population: All patients who received at least 1 dose of study drug.
Description: Baseline to the end of the study (Week 52)
Arm/Group | Indacaterol 300 μg Plus Placebo to Formoterol | Indacaterol 600 μg Plus Placebo to Formoterol | Formoterol 12 μg Plus Placebo to Indacaterol | Placebo to Indacaterol Plus Placebo to Formoterol
Serious Adverse Events (participants affected / at risk) | 63/437 | 51/425 | 69/434 | 48/432
Other Adverse Events (participants affected / at risk) | 199/437 | 183/425 | 164/434 | 176/432
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg Plus Placebo to Formoterol (N=437) | Indacaterol 600 μg Plus Placebo to Formoterol (N=425) | Formoterol 12 μg Plus Placebo to Indacaterol (N=434) | Placebo to Indacaterol Plus Placebo to Formoterol (N=432)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 3 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Microvascular angina (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Anterior capsule contraction (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 2 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 2
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 5 | 3
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0
Perianal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 5 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyothorax (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 4 | 0 | 5 | 4
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Laboratory test abnormal (Investigations) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 2 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18 | 12 | 32 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 1
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 2 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg Plus Placebo to Formoterol (N=437) | Indacaterol 600 μg Plus Placebo to Formoterol (N=425) | Formoterol 12 μg Plus Placebo to Indacaterol (N=434) | Placebo to Indacaterol Plus Placebo to Formoterol (N=432)
Lower respiratory tract infection (Infections and infestations) | 25 | 21 | 17 | 20
Nasopharyngitis (Infections and infestations) | 73 | 80 | 62 | 56
Upper respiratory tract infection bacterial (Infections and infestations) | 26 | 25 | 20 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 25 | 12 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 128 | 108 | 112 | 138
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 27 | 17 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.